CLINICAL TRIAL: NCT00618423
Title: The Effect of Perioperative Intravenous Low-dose Ketamine on Acute and Chronic Neuropathic Pain After Major Back Surgery. A Randomised, Placebo-controlled, Double-blind Study
Brief Title: The Effect of Perioperative Ketamine on Acute and Chronic Pain After Major Back Surgery
Acronym: KetaDol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christoph Czarnetzki, Responsable Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NAC 07-023 (07-006); Swissmedic 2007 DR 2198 (Other: Swiss Agency for Therapeutic products)
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Postoperative Pain
Keywords: Neuropathic pain; Chronic pain; Acute postoperative pain; Ketamine; Back surgery; Anesthesia; Perioperative
MeSH Terms: conditions — Pain, Postoperative; Neuralgia; Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiologic saline (Placebo Comparator)
  Interventions: Drug: Placebo
- Ketamine (Active Comparator)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Placebo — 50 ml syringes provided by the HUG pharmacy will contain 1% ketamine or 0.9% NaCl. After induction and before start of surgery, patients will receive an intravenous bolus of 0.025 ml/kg of the study solution (corresponding to 0.25 mg/kg ketamine). Maintenance will be with a syringe driver at a rate of 0.025 ml/kg/h (corresponding to 0.25 mg/kg/h ketamine) until one hour before the end of surgery, and will then be decreased to a rate of 0.01 ml/kg/h (corresponding to 0.1 mg/kg/h ketamine) throughout the stay in the recovery room (usually 2 to 3 hours). The infusion will be stopped when the patient leaves the recovery room.
  Arms: Physiologic saline
Drug: Ketamine — 50 ml syringes provided by the HUG pharmacy will contain 1% ketamine or 0.9% NaCl. After induction and before start of surgery, patients will receive an intravenous bolus of 0.025 ml/kg of the study solution (corresponding to 0.25 mg/kg ketamine). Maintenance will be with a syringe driver at a rate of 0.025 ml/kg/h (corresponding to 0.25 mg/kg/h ketamine) until one hour before the end of surgery, and will then be decreased to a rate of 0.01 ml/kg/h (corresponding to 0.1 mg/kg/h ketamine) throughout the stay in the recovery room (usually 2 to 3 hours). The infusion will be stopped when the patient leaves the recovery room.
  Other Names: Ketalar®
  Arms: Ketamine

SUMMARY:
After a surgical operation, patients may suffer from chronic pain. Ketamine, a well known anesthetic acts on receptors in the spine (NMDA receptors), which are implied in the occurrence of chronic pain. The mechanism is called central sensation. It is known that Ketamine reduces immediate postoperative pain, but its effectiveness in the prevention of the chronic pain is still unknown. The investigators study will follow patients until one year after operation for the occurrence of chronic pain. The investigators hypothesis is that Ketamine reduces significantly chronic postoperative pain after major back surgery and improves patient outcome.

There may be important inter-individual differences how persons react on a drug. These differences are partly determined by the genes of each individual. The investigators study includes therefore a genetic analysis.

Psychological and social factors also influence the perception of pain. It is still not well understood who these "psychosocial factors" determine the appearance and perception of chronic pain. In the investigators study the investigators will therefore study these factors by questionnaires.

DETAILED DESCRIPTION:
Background

1. Ketamine as an adjuvant to multimodal postoperative analgesia and its impact on the development of chronic neuropathic pain:

   Ketamine, a phenylcyclidine derivate, was developed in the 1960's to be used as a general anesthetic. The pharmacological mechanism of ketamine remained unclear for a long time. However, more recently, the antagonistic role of ketamine at the N-methyl-D-aspartate (NMDA) receptor was identified. Consequently, it has been suggested that ketamine should be used as an adjuvant for multimodal pain treatment.

   During the last 15 years, a large number of clinical trials have been published that tested ketamine for the management of acute postoperative pain. Three meta-analyses have confirmed an opioid sparing effect in the immediate postoperative period, a decrease in post-operative pain intensity, and an increase in the delay until the first request of rescue analgesia in patients who were randomised to intraoperative ketamine [Elia & Tramèr, 2005; Bell et al, 2005; Himmelseher & Durieux, 2005]. There was no evidence of an increase in the incidence of nightmares or unpleasant dreams when patients received low-dose ketamine as an adjuvant to a general anesthetic [Elia & Tramèr, 2005].

   Additionally to these short-term perioperative effects, ketamine is supposed to reduce the development of chronic neuropathic postoperative pain through NMDA receptor blockade and a reduction of wind-up and central sensitization [Woolf 2000]. Chronic postoperative pain is a major source of morbidity [Perkins & Kehlet, 2000]. Certain types of surgery, such as breast surgery, thoracotomy, inguinal hernia repair and limb amputation are considered as "high risk" interventions for developing neuropathic pain. After thoracotomy, for instance, incidences of chronic neuropathic pain up to 60% have been reported. A few studies only have looked at long-term outcomes. In a small pilot study, a beneficial effect of ketamine on persistent painful sensations around the scar was observed for up to 6 months after surgery [De Kock et al, 2001]. Chronic neuropathic pain remains an important therapeutic challenge. The pathophysiology of neuropathic pain has shown that central sensitisation might play an important role through hyperactivity/ hyperexcitability of spinal/supraspinal nociceptive neurons. Ketamine, which modulates NMDA receptors, is known to reduce neuropathic pain and might even prevent it. Furthermore, opioid resistance of neuropathic pain is a common feature and thermal sensory deficits within the painful area are predictive of the intensity of opioid response.

   In order to improve our understanding of the frequently observed variability in the response rate to ketamine, and to describe in more details the low back pain cohort we intend to study, we will address two further issues; first, pharmacogenetics of ketamine, and second, psychosocial factors that may influence the perception of postoperative pain and may predict the response to ketamine in patients with or without chronic low back pain.
2. Pharmacogenetics of ketamine:

   Factors that can affect the individual response to drugs are genetic and non-genetic, as for instance, compliance, age, body fat, nutrition, concomitant disease (such as liver and kidney diseases), and drugs or toxic substances (such as tobacco, alcohol, and environmental pollutants). The individual response to a drug is influenced by the combination of pharmacokinetic (absorption, distribution, metabolism, excretion) and pharmacodynamic processes. Each of these processes, as well as the underlying pathological painful condition, involves genetic and environmental factors that can affect the response to an analgesic. The only consistent and predictable factor might possibly be the genetic one, and thus pharmacogenetics may help individualizing drug treatment in accordance with the genetic "make-up" of the patient. Pharmacogenetic tests are now available in clinical practice and might help to better identify the best analgesic and also to estimate the optimal dose for an individual patient. Finally, this genetic knowledge should lead to mechanism-based approaches for the discovery of new analgesics.

   Polymorphic drug metabolizing enzymes and drug transporters affect the pharmacokinetics of drugs whereas polymorphic drug targets and disease related pathways influence the pharmacodynamic action of drugs [Samer et al, 2006]. Prospective trials are urgently needed to study the inherited susceptibility that may lead to a lack of therapeutic analgesic efficacy, or dose-dependent induced adverse drug reactions.

   We choose high-priority candidate polymorphisms that we predicted would be associated with pain-related response or resistance to post-operative pain treatment. CYP2C9, CYP3A4, CYP2D6 are alleles involved in the metabolism of analgesics such as non-steroidal anti-inflammatory drugs (NSAID), ketamine, tramadol, or ondansetron (for review, see [Samer et al, 2006]). As for pain sensitivity and morphine response variability, the met allele at the val158met polymorphisms in the catechol-O-methyltransferase gene (COMT), reduces the ability of the enzyme to metabolize catecholamines, and has been associated with a decrease in opioid consumption in cancer pain patients. Furthermore, COMT polymorphisms interacts with the nociceptive and emotional system since the variability in experimentally evoked pain thresholds is linked to this genetic polymorphisms [Zubieta et al, 2003]. Unpleasant pain-related affect, and anxiety disorders have also been associated with this polymorphisms [Olsson et al, 2005]. The met allele has been associated with depression and anxious temperament; both are well known risk factors for developing chronic pain [Hwang et al, 2005]. In addition to the a priori selection of these putative genes, we will carry out exploratory analyzes of polymorphisms in some additional genes that we had previously genotype for pain genetics studies. We recognize that correction for multiple testing might need a cohort of several hundred patients; thus, our observations and analyzes may be suitable only for generating hypotheses for future studies.
3. Psychosocial factors of pain perception in patients with back pain undergoing surgery:

Pain intensity is strongly associated with disability. Aside the importance of symptoms, function, general well-being, work status, and satisfaction with care have been proposed as a core set of outcomes in clinical trials and routine care settings [Mannion et al, 2005]. Psychological distress and depressive mood increase the risk of chronicity. A systematic review evaluated psychological predictors of chronicity and disability in prospective cohorts of low back pain patients [Pincus et al, 2002]. Increased risk of chronicity (i.e. persisting symptoms and/or disability) as a result of psychological distress and depressive mood emerged as the main finding.

Patients' beliefs and expectations about their pain problem also seem to influence the recovery process. Patients' expectations about treatment have been shown to influence the outcome, i.e. functional improvement, for example, can be linked not only to the intrinsical value of treatment but also to the patients' expectations of its possible benefits. Lutz et al showed that patients with higher expectations of surgery had better outcomes than those with lower expectations [Lutz et al, 1999]. Iversen et al found that patients with many preoperative expectations tended to improve more than those with fewer expectations [Iversen et al, 1998]. More ambitious expectations for physical function were also associated with improved function and satisfaction with physical function; however, high expectations for pain relief were associated with greater report of pain and decreased satisfaction with pain relief, thus suggesting that these types of expectations should be addressed differently in preoperative discussions.

Investigating the relationship between expected results and actual outcomes, McGregor & Hughes assessed patients' expectations of surgery, and satisfaction with outcome in terms of pain, function, disability and general health at 6 weeks, 6 months and 1 year [McGregor & Hughes, 2002]. The results showed that patients had high expectations of recovery and were confident of achieving this recovery. As for satisfaction, however, patients' reports at all review stages indicated that surgery had achieved only part of what they had expected, suggesting that patients had unrealistic expectations leading to lower satisfaction levels.

Painful experiences may be accompanied by catastrophizing cognitions, i.e. pessimistic beliefs and expectations regarding the self, the others and the future, which may give rise to feelings of helplessness concerning one's ability to cope with life events. This may lead to pain-related fear, avoidance behaviors, and to reduced activity. Disability and disuse may ensue and be associated with depression, thus increasing pain and catastrophizing and setting into motion a vicious circle. When back pain is not associated with catastrophizing thoughts, the absence of fear allows for the confrontation with activity and eventually for recovery [Vlaeyen & Linton, 2000]. This model refers to both cognitive factors (e.g. meaning of pain, expectations regarding control over pain, maladaptive thoughts) and behavioural responses that may be active (e.g. carrying on with daily activities, exercising) or passive (e.g. rest, giving up control, withdrawal from activities) [Picavet et al, 2002].

ELIGIBILITY:
Inclusion Criteria:

* Adults, age ≥18 years, male or female
* American Society of Anaesthesiology (ASA) status I-III.
* Back surgery: laminectomy, lumbar arthrodesis (Posterior Lumbar Interbody Fusion - PLIF, Transforaminal Lumbar Interboby Fusion - TLIF, Postero-lateral Fusion, semi-rigid fixation).
* Subjects who have signed and dated an informed consent to participate in the study during the pre-operative assessment.

Exclusion Criteria:

* Coronary heart disease (unstable angina, MI within the last 6 months)
* Glaucoma.
* History of allergy or hypersensitivity to ketamine or morphine.
* Dementia or inability to understand the study protocol.
* Subjects who have taken any investigational drug or used an experimental medical device within 30 days before the start of the study or are currently enrolled in another investigational drug study.
* Failed back surgery syndrome (i.e. an unfavourable condition of a patient following back or spine surgery).
* Posttraumatic paraplegia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the long-term (6 and 12 months) effect of perioperative intravenous low-dose ketamine on chronic neuropathic pain in patients undergoing major back surgery. | one year

SECONDARY OUTCOMES:
To evaluate the short-term (during hospitalisation) effect of perioperative intravenous low-dose ketamine in patients undergoing major back surgery: tolerability and safety, opioid-sparing effect, pain intensity, morphine-related adverse effects. | one week
To study the potential impact of genetic variability of several enzymes (CYP2D6, CYP2C9, COMT) known to modulate pain sensitivity and/or metabolism of opioid and NSAIDs on analgesic consumption and ketamine response. | immediate
To study psychosocial factors that may be involved in the perception of acute and chronic postoperative pain in patients with or without chronic back pain undergoing back surgery. | one year
To study the pharmakokinetics of an intravenous low-dose ketamine infusion. | one day

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tramèr, Prof, MD, PhD, Study Chair — anesthesia department; Christoph A Czarnetzki, MD, MBA, Principal Investigator — anesthesia department
Locations (1):
- University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Czarnetzki C, Desmeules J, Tessitore E, Faundez A, Chabert J, Daali Y, Fournier R, Dupuis-Lozeron E, Cedraschi C, Richard Tramer M. Perioperative intravenous low-dose ketamine for neuropathic pain after major lower back surgery: A randomized, placebo-controlled study. Eur J Pain. 2020 Mar;24(3):555-567. doi: 10.1002/ejp.1507. Epub 2019 Dec 9. PMID 31743533